CLINICAL TRIAL: NCT01678391
Title: Feasibility of Endoscopic Ultrasound Based Biliary Stone Removal Without Fluoroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: University of California, Los Angeles (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Janak Shah, MD, Director of Pancreatic and Biliary Endoscopy, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012.065-1
Record Dates: First submitted 2012-08-29; First posted 2012-09-05 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Common Bile Duct Gall Stones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with common bile duct stones. (Experimental): Common bile duct stone removal without fluoroscopy
  Interventions: Procedure: Common bile duct stone removal without fluoroscopy.

INTERVENTIONS:
Procedure: Common bile duct stone removal without fluoroscopy. — ERCP stone extraction technique without fluoroscopy involves: (1) catheter or catheter with wire access into the bile duct, (2) confirmation of biliary access with catheter aspiration of bile, (3) performance of endoscopic biliary sphincterotomy or balloon dilation to widen the bile duct opening to permit stone removal, (4) stone removal - number of stones seen on EUS should match the number removed.

SUMMARY:
To assess the feasibility and success of endoscopic ultrasound (EUS) directed biliary stone removal without use of fluoroscopy. Success for this study will be defined as the successful removal of all stones from the bile duct without the use of fluoroscopy. Fluoroscopy will only be used at the end of a presumed successful procedure to confirm that all stones are removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients able to give informed consent
* Patients referred to IES for the endoscopic evaluation and treatment of suspected bile duct stones

Exclusion Criteria:

* Patients with >3 bile duct stones or with any stone >12mm on EUS
* Patients with no bile duct stones on EUS
* Patients with altered biliary anatomy (periampullary diverticulum, anomalous pancreatibiliary junction, altered surgical anatomy)
* Patients who are pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Successful removal of all stones from the bile duct without the use of fluoroscopy. | Up to 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Janak Shah, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center, San Francisco, California, United States

REFERENCES:
- [Background] Carr-Locke DL. Overview of the role of ERCP in the management of diseases of the biliary tract and the pancreas. Gastrointest Endosc. 2002 Dec;56(6 Suppl):S157-60. doi: 10.1067/mge.2002.129023. No abstract available. PMID 12447259
- [Background] Shelton J, Linder JD, Rivera-Alsina ME, Tarnasky PR. Commitment, confirmation, and clearance: new techniques for nonradiation ERCP during pregnancy (with videos). Gastrointest Endosc. 2008 Feb;67(2):364-8. doi: 10.1016/j.gie.2007.09.036. PMID 18226705
- [Background] Menees S, Elta G. Endoscopic retrograde cholangiopancreatography during pregnancy. Gastrointest Endosc Clin N Am. 2006 Jan;16(1):41-57. doi: 10.1016/j.giec.2006.01.004. PMID 16546022
- [Derived] Shah JN, Bhat YM, Hamerski CM, Kane SD, Binmoeller KF. Feasibility of nonradiation EUS-based ERCP in patients with uncomplicated choledocholithiasis (with video). Gastrointest Endosc. 2016 Nov;84(5):764-769. doi: 10.1016/j.gie.2016.03.1485. Epub 2016 Mar 31. PMID 27040099